CLINICAL TRIAL: NCT01295476
Title: Biological Correlates With T-cell Acute Lymphoblastic Leukemia (T-ALL) Gene Expression and Clinical Outcome
Brief Title: Biomarker Study in Bone Marrow Samples From Patients With T-Cell Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL10B1; COG-AALL10B1; CDR0000695252; AALL10B1 (Other: COG); NCI-2011-02848 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Gene Expression Profiling; Microarray Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone Marrow

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in bone marrow samples from patients with T-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To confirm an association between induction failure (IF) status predicted by a previously identified 116-member genomic classifier and actual induction therapy outcome observed on COG study AALL0434.
* To explore whether there is an association between early relapse (as defined by bone marrow or extramedullary relapse within 18 months of diagnosis) predicted by previously identified 5-member (primary) and 57-member (secondary) genomic classifiers, and actual relapse status at 18 months on COG study AALL0434. (Exploratory)

OUTLINE: RNA from cryopreserved bone marrow samples are analyzed for gene expression by microarray methods. Samples are then compared with the 116-member genomic classifier.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed T-cell acute lymphoblastic leukemia
* Cryopreserved bone marrow from the Children Oncology Group (COG) Cell Bank of patients enrolled on COG-AALL03B1 and COG-AALL0434, including the following:

  * 30 samples from patients who had > 25% bone marrow blasts at day 29 (induction failure [IF] cases)
  * Samples of cases of bone marrow and/or CNS relapse occurring within the first 18 months of treatment
  * Random samples of 105 non-IF cases who achieved remission at the end of induction therapy (at least 18 months)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newly diagnosed T-cell acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Association between induction failure status predicted by 116-member genomic classifier and actual induction therapy outcome observed on COG study AALL0434

CONTACTS AND LOCATIONS:
Overall Officials: Stuart S. Winter, MD, Principal Investigator — University of New Mexico Cancer Center